CLINICAL TRIAL: NCT00495443
Title: Peterio™ - an Add-on Device for Enhanced Safety of Aesthetic Laser Treatments
Brief Title: Enhanced Safety Aesthetic Laser System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Scilex Ltd. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Peterio-06
Record Dates: First submitted 2007-07-01; First posted 2007-07-03 (Estimated); Last update posted 2007-07-03 (Estimated); Status verified 2007-07

CONDITIONS: Hirsutism; Hypertrichosis; Telangiectases; Rhytides
MeSH Terms: conditions — Hirsutism; Hypertrichosis; Telangiectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Peterio

SUMMARY:
The purpose of this study is to determine whether a new laser system provides better safety and efficacy than existing lasers in popular cosmetic procedures such as hair removal, treatment of cosmetically disturbing vascular lesions and rhytides.

DETAILED DESCRIPTION:
Cosmetic lasers are a well-established, popular modality for removal of unwanted hair, treatment of all types of vascular lesions, including hemangiomas, port wine stains, and a variety of telangiectases as well as facial rhytides reduction. The existing lasers are based on a wavelength that is specifically absorbed by the chromophore found in the target such as hair follicle, where the energy is converted to heat resulting in a thermal injury. However, the lasers for cosmetic treatments are not without limitations. A laser based long-term hair removal treatment is based on thermal destruction of the hair shaft and follicle using wavelengths that are specifically absorbed by the pigment melanin found in the hair follicle. The heating of hair follicle is done through heat dissipation from the hair shaft. One of the significant limitations of this approach is the fact that the epidermis through which the light energy must penetrate is rich in melanin and therefore absorbs a major portion of the energy, resulting in inadequate heating of the hair follicles. Similar problem exists when targeting other chromophores such as hemoglobin or water. The purpose of the study is an evaluation of safety and efficacy of a new laser based device.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years old
* Fitzpatrick skin types I to VI
* Unwanted hair or/and
* Aesthetically disturbing vascular lesions or/and
* Facial rhytides

Exclusion Criteria:

* Age below 18 or above 75 year old.
* Use of photosensitive medications
* Photosensitive diseases
* Active infection of any type and active infection or or a history of Herpes Simplex in the treated site
* Exposure to sun or artificial tanning during the last 3-4 weeks
* For treatment of facial rhytides- surgical or nonsurgical facial procedure (i.e., laser skin resurfacing, dermabrasion, phenol peel, nonablative laser, or temporary/permanent filler (e.g., collagen, fat, hyaluronic acid injections)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2007-09; Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
Hair, vascular lesions and wrinkles reduction as counted 1-3 months after each treatment session, depending on the treated area.

SECONDARY OUTCOMES:
Measuring treatment discomfort as graded by the patients

CONTACTS AND LOCATIONS:
Overall Officials: Leon Gilad, MD, Principal Investigator — Hadassah Medical Center, Dermatology
Locations (1):
- Hadassah Medical Center, Dermatology, Jerusalem, Israel

REFERENCES:
- [Background] Anderson RR, Parrish JA. Selective photothermolysis: precise microsurgery by selective absorption of pulsed radiation. Science. 1983 Apr 29;220(4596):524-7. doi: 10.1126/science.6836297.